CLINICAL TRIAL: NCT02694679
Title: Randomized Controlled Trial of Social Network Targeting to Magnify Population-Level MNCH Behavior Change in Honduras
Brief Title: Randomized Controlled Trial of Social Network Targeting in Honduras
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Inter-American Development Bank (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 1506016012
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Preterm Delivery; Hypothermia; Diarrhea; Upper Respiratory Infection; Omphalitis
Keywords: social networks, maternal and child health, global health
MeSH Terms: conditions — Premature Birth; Hypothermia; Diarrhea; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (16):
- Random 0 (No Intervention): The CBNH intervention will be delivered to 0% of population targeted households in the village.
- Random 5 (Active Comparator): The CBNH intervention will be delivered to a random 5% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Random 10 (Active Comparator): The CBNH intervention will be delivered to a random 10% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Random 20 (Active Comparator): The CBNH intervention will be delivered to a random 20% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Random 30 (Active Comparator): The CBNH intervention will be delivered to a random 30% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Random 50 (Active Comparator): The CBNH intervention will be delivered to a random 50% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Random 75 (Active Comparator): The CBNH intervention will be delivered to a random 75% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Random 100 (Active Comparator): The CBNH intervention will be delivered to a random 100% of targeted households in the village.
  Interventions: Behavioral: CBNH
- Friendship 0 (No Intervention): CBNH 0% of population targeted
- Friendship 5 (Experimental): The CBNH intervention will be delivered to 5% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH
- Friendship 10 (Experimental): The CBNH intervention will be delivered to 10% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH
- Friendship 20 (Experimental): The CBNH intervention will be delivered to 20% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH
- Friendship 30 (Experimental): The CBNH intervention will be delivered to 30% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH
- Friendship 50 (Experimental): The CBNH intervention will be delivered to 50% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH
- Friendship 75 (Experimental): The CBNH intervention will be delivered to 75% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH
- Friendship 100 (Experimental): The CBNH intervention will be delivered to 100% of households identified through friendship nomination.
  Interventions: Behavioral: CBNH

INTERVENTIONS:
Behavioral: CBNH — The household-level intervention package targets health behaviors surrounding neonatal and maternal health, and diarrhea and respiratory illness prevention and management.
  Arms: Friendship 10; Friendship 100; Friendship 20; Friendship 30; Friendship 5; Friendship 50; Friendship 75; Random 10; Random 100; Random 20; Random 30; Random 5; Random 50; Random 75

SUMMARY:
Social network targeting strategies can be used to improve the delivery and uptake of health interventions. We will enroll approximately 30,000 individuals into a randomized controlled trial of different targeting algorithms in order to explore how social network dynamics affect the uptake, diffusion, and group-level normative reinforcement of key neonatal and infant health behaviors and attitudes in 176 rural villages in the Copan region of Honduras. Our goal is to develop methods by which global health practitioners can exploit face-to-face social network interactions in order to maximize uptake of neonatal and infant health interventions. The villages will be randomly assigned to 16 cells of 11 villages each in a 2 x 8 factorial design of different targeting algorithms.

DETAILED DESCRIPTION:
Honduras has one of the highest neonatal mortality rates in Latin America despite having made significant strides in reducing neonatal, infant, and child mortality in the last several decades. Although many neonatal and infant deaths can be prevented through provision of clinical care services, emerging evidence also suggests that a substantial reduction in neonatal and infant mortality can also be achieved with simple, low-cost interventions within family and community settings. This is particularly important in areas where functional community health facilities are not available. Family and community outreach programs can serve to educate families about beneficial home care practices.

In order to accelerate neonatal mortality reduction , there is an urgent need to develop innovative solutions that are not only effective, but also more easily implementable and more readily scalable. An important component of this challenge, which has hitherto not been effectively measured and understood with respect to neonatal mortality, is the "embeddedness" of individuals within social networks. Hence, through a large-scale randomized controlled trial (RCT) in rural Honduras, we will deploy and assess social network targeting algorithms in order to maximize diffusion and adoption of the "Changing behaviors to improve neonatal, child, and maternal health using communication and social networks at the community level intervention (CBNH)". The CBNH intervention is a household-level intervention package that targets health behaviors surrounding neonatal and maternal health, and diarrhea and respiratory illness prevention and management implemented by the Inter-American Development Bank (IADB) and their partners.

This RCT is aimed at discerning optimal methods for targeting delivery of the intervention to the population. Specifically we will (1) test what percentage of a community needs to be in a program to achieve social norms change around key neonatal care behaviors, and (2) test whether so-called nominated-friend-targeting, a method that targets individuals who are more highly connected in the network, is more effective than a control strategy. Our 2x8 factorial design will examine how large a subset of the population should be used as a "seed" group in order to maximize the chances of spread of the effect, and the efficiency with which such an intervention might be delivered in the future. To do this, we will assign each of the 176 study villages to either one of the two groups: 1)random assignment (active comparator), where "seed" individuals are chose at random or 2) friend-of-random assignment (experimental), where "seed" individuals are chosen on the basis of being named as a friend of a randomly selected individual. Each of the groups of villages will also be assigned to one of eight treatment percentages (0%, 5%, 10%, 20%, 30% 50%, 75%, 100%), where each represents the percent of targeted households in that village to receive the CBNH health intervention.

ELIGIBILITY:
Inclusion Criteria: People who live or work in target villages, ages 12 and up -

Exclusion Criteria: People who do not live or work in the sample villages, and those who are prisoners, mentally impaired, or under age 12 years.

-

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31195 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Speed of adoption of intervention and fraction of adoption of CBNH intervention (participant survey). | 24 Months
Percent of participants reporting paternal involvement during pregnancy and postpartum care (participant survey). | 24 Months
Percent of newborns with appropriate umbilical cord care (participant survey) | 24 Months
Percent of children under 5 with diarrheal illness in the last 4 weeks (participant survey) | 24 Months
Percent of children under age 5 with symptoms of acute respiratory illness in the last 4 weeks (participant survey). | 24 months
Percent of women experiencing a pregnancy danger sign who sought professional medical care (participant survey). | 24 months
Percent of children experiencing a newborn danger sign who were taken to professional medical care (participant survey) | 24 months
Percent of children who were breastfed exclusively during first 6 months (participant survey) | 24 Months
Percentage of deliveries taking place in medical facilities (participant survey, medical records). | 24 months
Receipt of post-natal care medical check-up within 7 days of delivery - Mother (participant survey, medical records). | 24 months
Receipt of post-natal care medical check-up within 7 days of delivery - Newborn (participant survey, medical records). | 24 months
Percent of newborns receiving appropriate thermal care during first 7 days after birth (participant survey). | 24 months

SECONDARY OUTCOMES:
Knowledge/attitudes about thermal care in newborns (Participant survey) | 24 months
Knowledge/attitudes about paternal involvement (Participant survey) | 24 months
Knowledge/attitudes about proper cord care (Participant survey) | 24 months
Knowledge/attitudes about prevention and/or treatment of diarrhea (Participant survey) | 24 months
Knowledge/attitudes about prevention and/or treatment of respiratory illness (Participant survey) | 24 months
Knowledge about danger signs during pregnancy (Participant survey). | 24 months
Knowledge about danger signs for newborns (Participant survey). | 24 months
Knowledge/attitudes about facility-based births (Participant survey). | 24 months
Knowledge/attitudes about post-natal care for women (Participant survey). | 24 months
Knowledge/attitudes about post-natal care for newborns (Participant survey). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Christakis, MD, PhD, Principal Investigator — Yale University
Locations (2):
- Yale Institute for Network Science, New Haven, Connecticut, United States
- Community intervention, Copán, Copán Department, Honduras

REFERENCES:
- [Background] Shakya HB, Stafford D, Hughes DA, Keegan T, Negron R, Broome J, McKnight M, Nicoll L, Nelson J, Iriarte E, Ordonez M, Airoldi E, Fowler JH, Christakis NA. Exploiting social influence to magnify population-level behaviour change in maternal and child health: study protocol for a randomised controlled trial of network targeting algorithms in rural Honduras. BMJ Open. 2017 Mar 13;7(3):e012996. doi: 10.1136/bmjopen-2016-012996. PMID 28289044
- [Derived] Oles W, Alexander M, Negron R, Nelson J, Iriarte E, Airoldi EM, Christakis NA, Forastiere L. Maternal and child health intervention to promote behaviour change: a population-level cluster-randomised controlled trial in Honduras. BMJ Open. 2024 Jun 10;14(6):e060784. doi: 10.1136/bmjopen-2022-060784. PMID 38858139